CLINICAL TRIAL: NCT03148158
Title: Assessment Of Bladder Tumors Stage And Grade By Outpatient Flexible Cystoscopy Performed By Urology Resident
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Urology Msc, Oncology fellow at Urology and Nephrology Center, Principal Investigator, Mansoura University
Other Study IDs: F-Cystoscopy NMIBC
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-05

CONDITIONS: Bladder Cancer; Flexible Cystoscopy; Non-muscle Invasive Bladder Cancer (NMIBC); Pain, Postoperative
Keywords: Bladder Cancer; Flexible cystoscopy; Diagnosis
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Pain, Postoperative; Disease | interventions — Cystoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bladder biopsy and urine cytology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cystoscopy — Outpatient flexible cystoscopy and inpatient rigid cystoscopy

SUMMARY:
This will be a prospective trial comparing the perspective gross morphological of bladder tumor assessment done by outpatient flexible cystoscopy performed by resident, inpatient rigid cystoscopy done by senior staff and their prediction of the degree of invasion of bladder tumor plus the prediction of the grade compared with the standard pathological result.

Also, assessment of the patient reported outcomes after both flexible and rigid cystoscopy will be done.

In the long run of the study, the prognostic gross morphology with recurrence, progression and cancer specific survival will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years or older
* Denovo or recurrent NMIBC
* Bladder mass discovered in hematuria investigation
* Willing to share in study

Exclusion Criteria:

* inability to cooperate with flexible cystoscopic evaluations
* cystoscopies for other kind of intervention (e.g., removal of a ureteral stent)
* Untreated infections
* Other causes of storage or voiding symptoms as untreated benign prostatic hyperplasia (BPH) or interstitial cystitis
* Unpassable urethral stricture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with suspected denovo, recurrent bladder mass or hematuria needing assessment by flexible cystoscopy will be asked to participate in this study at Urology and Nephrology Center Outpatient Clinics and will be provided with an informed consent form in line with Good Clinical Practise and the Declaration of Helsinki.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of clinical grade and stage of bladder lesions diagnosed by flexible cystoscopy done by urology residents | 1 year
  Outcome measures by histopathological results of bladder biopsy

SECONDARY OUTCOMES:
Evaluation of pain perception in patient undergoing flexible or rigid diagnostic cystoscopy | 1 year
  Outcome measures by visual analog scale (VAS) pain score
Assessment of the patient reported outcomes after both flexible and rigid cystoscopy | 1 year
  Outcome measures by Freiburg Index of Patient Satisfaction (FIPS) questionnaire
Assessment of the prognostic value of gross morphology with recurrence, progression | 2 year
  Outcome measures by Number of patients surviving for two year without tumor recurrence will be counted and compared

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Abol-Enein, MD, Study Chair — Urology and Nephrology center; Ahmed Mosbah, MD, Study Director — Urology and Nephrology center; Mohamed Abdelbaset, Msc, Principal Investigator — Urology and Nephrology Center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
meta-analyses by contact the Prof. Hassan Abol-Enein, MD, Phd (Study Chair)